CLINICAL TRIAL: NCT06914583
Title: A Prospective, Multi-center, Randomized, No-treatment Controlled, Evaluator-blinded, Superiority Clinical Trial to Evaluate the Safety and Effectiveness of Sodium Hyaluronate 32 mg/ml for Improvement of Facial Skin Dryness and Dullness
Brief Title: Safety and Efficacy Evaluation of Sodium Hyaluronate 32mg/ml in Improving Facial Skin Dryness and Dullness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IBSA Farmaceutici Italia Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23CHN-Pro-IT01
Record Dates: First submitted 2025-03-17; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Facial Dryness; Facial Dullness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Experimental): The treatment group will receive intradermal injections of sodium hyaluronate
  Interventions: Device: Sodium Hyaluronate
- Control group (No Intervention): The control group will not receive any treatment

INTERVENTIONS:
Device: Sodium Hyaluronate — Sodium Hyaluronate 32 mg/ml
  Arms: Treatment group

SUMMARY:
The aim of the study is to evaluate the safety and efficacy of sodium hyaluronate 32 mg/ml in improving facial skin dryness and dullness. Subjects are randomized to the treatment group or to the control group. Only subjects in the treatment group are treated by intradermal injection.

DETAILED DESCRIPTION:
This is a prospective multi-center clinical investigation. Enrolled subjects are randomized to the treatment group or to the no-treatment control group. The treatment group will receive intradermal injections of sodium hyaluronate 32 mg/ml. The improvement of facial skin dryness and dullness will be evaluated at multiple timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and ≤65 years old (based on the time of signing the ICF), gender is not restricted;
2. Skin Fitzpatrick is classified as type II-IV;
3. Subjects who are seeking temporary improvement of their dry facial skin and dull complexion. The investigator has assessed the subjects are suitable for receiving injectable treatment to improve these conditions;
4. Subjects who have agreed not to use any other medical cosmetic treatments related to the study during the study period;
5. Subjects who voluntarily sign a written informed consent form, and able to comprehend the full nature and the purpose of the investigation, including possible risks and side effects, and subjects able to cooperate with the investigator and to comply with the requirements of the entire investigation (including ability to attend all the planned investigation visits according to the time limits), based on investigator's judgement.

Exclusion Criteria:

1. Known allergy to hyaluronic acid or any component of this product;
2. Known history of severe allergies;
3. Known history of severe autoimmune disease;
4. Subjects with episode of herpes cutis;
5. Subjects with cicatricial diathesis;
6. Facial area has unknown injection substances;
7. Have received any permanent or semi-permanent fillers at the facial area (e.g., calcium hydroxyapatite, poly-L-lactic acid, polymethyl methacrylate, silicones, expanded polytetrafluoroethylene (ePTFE), polycaprolactone, etc.), autologous fat, face lift (including thread lifts), etc., or plan to receive any of the above treatments during the investigation;
8. Have received temporary dermal filler treatment (e.g., cross-linked hyaluronic acid, collagen) at the facial area within the 12 months prior to enrolment, or plan to receive any of the above treatments during the investigation;
9. Have received botulinum toxin injection, mesotherapy, or facial cosmetic procedures (e.g., facial liposuction, cosmetic surgery, face slimming, photo modulation therapy, intense pulsed light, radiofrequency, non-cross-linked hyaluronic acid injection (except for mesotherapy), dermabrasion, laser or chemical peels or other ablation procedures, etc.) at facial area within 6 months prior to enrolment, or plan to receive any of the above treatments during the investigation;
10. Have received sodium hyaluronate compound solution injection (mesotherapy, etc) at facial area within 3 months prior to enrolment,
11. Facial area has active or progressive skin infection (including viral, bacterial, fungal);
12. Facial area has skin granuloma;
13. Facial area has active or progressive skin diseases or with isomorphic reactions such as acute eczema, flat warts, lichen planus, psoriasis vulgaris, etc.;
14. Facial area has malignant tumors or skin tumors of unknown nature;
15. Subjects who work outdoors for a long time or need to be exposed to sunlight after surgery;
16. Patients with excessive expectations for treatment effects;
17. Subjects with coagulation dysfunction or other systemic diseases;
18. Subjects undergoing chemotherapy/radiotherapy;
19. Subjects with mental illness or emotional instability;
20. Subjects who had received any thrombolytic agents, anticoagulants or antiplatelet drugs within 2 weeks before enrolment;
21. Subjects who are pregnant or planned to become pregnant during the investigation period, or breastfeeding;
22. Subject who participated in other clinical investigation within 1 month prior to enrolment in this investigation, or currently participating in other clinical investigation;
23. The investigator considers that the subject is not suitable to participate in this clinical investigation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
GAIS (Global Aesthetic Improvement Scale) - Blinded evaluator | 12 week
  Treatment effective rate (third-party blinded investigator assessment)

SECONDARY OUTCOMES:
GAIS-Blinded evaluator | 4week, 8week, 10week, 16week, 20week
  Treatment effective rate (third-party blinded investigator assessment)
GAIS-Investigator | 4week, 8week, 10week, 12week, 16week, 20week
  Treatment effective rate (treating investigator assessment)
GAIS-Subject | 4week, 8week, 10week, 12week, 16week, 20week
  Treatment effective rate (subject assessment)
Improvement of skin moisture | 4week, 8week, 10week, 12week, 16week, 20week
  Corneometer assessment
Skin dryness improvement assessment - Investigator | 4week, 8week, 10week, 12week, 16week, 20week
  Dryness improvement assessment will be performed by the treating investigator. The following scoring will be applied: -1: worse, 0= no change, 1=improvement.
Skin dryness improvement assessment - Subject | 4week, 8week, 10week, 12week, 16week, 20week
  Dryness improvement assessment will be performed by the subect. The following scoring will be applied: -1: worse, 0= no change, 1=improvement.
Skin dullness improvement assessment - Investigator | 4week, 8week, 10week, 12week, 16week, 20week
  Skin dullness improvement assessment will be performed by the treating investigator. The following scoring will be applied: -1: worse, 0= no change, 1=improvement.
Skin dulless improvement - Subject | 4week, 8week, 10week, 12week, 16week, 20week
  Skin dullness improvement assessment will be performed by the subject. The following scoring will be applied: -1: worse, 0= no change, 1=improvement.
Subject treatment satisfaction assessment scale | 4week, 8week, 10week, 12week, 16week, 20week
  For the question "How do you feel satisfied with the treatment effect of the investigational product?", the answer criteria are from 1 to 5, where 1= very dissatisfied and 5= very much satisfied.
Red blood cell (RBC) | 0week, 12week, 32 week
White blood cell (WBC) | 0week, 12week, 32 week
Platelet count (PLT) | 0week, 12week, 32 week
Hemoglobin (HGB) | 0week, 12week, 32 week
Serum alanine aminotransferase (ALT) | 0week, 12week, 32 week
Serum aspartate aminotransferase (AST) | 0week, 12week, 32 week
Serum urea nitrogen/urea (BUN/Urea) | 0week, 12week, 32 week
Serum creatinin (Cr) | 0week, 12week, 32 week
Blood glucose (GLU) | 0week, 12week, 32 week
Urine pH | 0week, 12week, 32 week
Urine glucose | 0week, 12week, 32 week
Urine protein | 0week, 12week, 32 week
Urine specific gravity | 0week, 12week, 32 week
Urine red blood cell count | 0week, 12week, 32 week
Urine white blood cell count | 0week, 12week, 32 week
Urine nitrite | 0week, 12week, 32 week
Prothrombin time (PT) | 0week
Activated partial thromboplastin time (APTT) | 0week
Thrombin time (TT) | 0week
Fibrinogen (FIB) | 0week
Blood pressure (mmHg) | 0week, 4week, 8week, 10week, 12week, 16week, 20week, 32week
  Systolic blood pressure and diastolic blood pressure will be measured
Temperature (°C) | 0week, 4week, 8week, 10week, 12week, 16week, 20week, 32week
Respiration rate | 0week, 4week, 8week, 10week, 12week, 16week, 20week, 32week
  Times/min
Heart rate | 0week, 4week, 8week, 10week, 12week, 16week, 20week, 32week
  Beats/min
Incidence rate of adverse events (AEs) | 0week, 1week, 2week, 4week, 5week, 6week, 8week, 9week, 10week, 12week, 16week, 20week, 32week
  Incidence rate (%) and number of adverse events (AEs)
Incidence rate of serious adverse events (SAEs) | 0week, 1week, 2week, 4week, 5week, 6week, 8week, 9week, 10week, 12week, 16week, 20week, 32week
  Incidence rate (%) and number of serious adverse events (SAEs)
Incidence rate of adverse device effects (ADE) | 0week, 1week, 2week, 4week, 5week, 6week, 8week, 9week, 10week, 12week, 16week, 20week, 32week
  Incidence rate (%) and number of adverse device effects (ADE)
Incidence rate of serious adverse device effects (SADE) | 0week, 1week, 2week, 4week, 5week, 6week, 8week, 9week, 10week, 12week, 16week, 20week, 32week
  Incidence rate (%) and number of serious adverse device effects (SADE)
Incidence rate of injection site reactions | 1week, 2week, 4week, 5week, 6week, 8week, 9week, 10week
  Incidence rate (%) and number of injection site reactions
Incidence rate of device deficiencies | 0week, 4week, 8week
  Incidence rate (%) and number of of device deficiencies

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Peking Union Medical College Hospital (PUMCH), Beijing
  - Peking University First Hospital, Beijing
  - The First Principle Hospital of Changde City, Changde
  - West China Hospital of Stomatology Sichuan Hospital, Chengdu
  - Tongji Hospital of Tongji University, Shanghai
  - The Second Affiliated Hospital Of Xi'an Jiaotong University, Xi'an